CLINICAL TRIAL: NCT06685354
Title: Sequential Targeted and Immunotherapy With Recombined Human Type 5 Adenovirus Via Hepatic Arterial Infusion for BCLC Stage C Hepatocellular Carcinoma: A Prospective Single-Center Single-Arm Pilot Study
Brief Title: Sequential T and I With H101 Via HAI for BCLC C Stage HCC: A Prospective Single-Center Single-Arm Pilot Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-281-002
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): The participants will receive hepatic arterial infusion of recombinant human adenovirus type 5 injection in combination with first-line targeted and immunotherapy as recommended by the 2024 primary liver cancer treatment guidelines.
  Interventions: Drug: hepatic arterial infusion of recombinant human type 5 adenovirus

INTERVENTIONS:
Drug: hepatic arterial infusion of recombinant human type 5 adenovirus — Participants will receive hepatic arterial infusion of recombinant human type 5 adenovirus (H101). The H101 treatment regimen consists of 3 cycles or until a specific treatment discontinuation event occurs as outlined in the protocol. The H101 administration method is as follows: if the sum of the largest diameters of lesions is ≤10 cm, the total dose is 1.0×10^12 vp (2 vials); if the sum of the largest diameters is >10 cm, the total dose is 1.5×10^12 vp (3 vials). Treatment cycles are every 3 weeks.

SUMMARY:
Indication: Hepatocellular carcinoma (HCC) patients at Barcelona Clinic Liver Cancer (BCLC) stage C.

Study Objectives: This study aims to use a prospective single-center single-arm pilot approach to preliminarily obtain data on the recent efficacy and safety of sequential targeted and immunotherapy with recombinant human type 5 adenovirus (H101) administered via hepatic arterial infusion for BCLC stage C HCC. Additionally, it will explore changes in the patients' immune systems before and after treatment, providing a basis for formal research.

Study Content: The study will use a prospective single-center single-arm pilot design to preliminarily assess the efficacy of sequential targeted and immunotherapy with H101 via hepatic arterial infusion in BCLC stage C HCC. Primary efficacy endpoints include: Objective Response Rate (ORR). Secondary efficacy endpoints include: Disease Control Rate (DCR), Duration of Response (DOR), Progression-Free Survival (PFS) at 6 months and 12 months, Overall Survival (OS) at 6 months and 12 months, Median Progression-Free Survival (mPFS), Liver-specific PFS. Additionally, the study will collect data on safety and tolerability and will explore changes in peripheral blood lymphocytes before and after treatment.

Expected Objectives: Efficacy and Safety Assessment: To preliminarily gather data on the short-term efficacy, safety, and tolerability of sequential targeted and immunotherapy using hepatic arterial infusion of H101 in patients with BCLC stage C HCC. This includes assessing primary efficacy endpoints (e.g., objective response rate) and secondary efficacy endpoints (e.g., disease control rate, duration of response, progression-free survival, overall survival, etc.). Immune System Changes: To investigate the patterns of peripheral blood lymphocyte changes before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in the study, signing the informed consent form, and willing to undergo follow-up;
2. Age ≥ 18 years and ≤ 75 years, regardless of gender;
3. Clinically or pathologically confirmed BCLC Stage C hepatocellular carcinoma, with no prior TACE or systemic treatment;
4. Baseline imaging (MRI or CT) showing measurable lesions with a longest diameter ≥ 1 cm;
5. Child-Pugh score ≤ 7 (Child-Pugh A-B);
6. Liver tumor burden not exceeding 50% of the liver volume;
7. Able to swallow pills normally;
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 (see Appendix 1 for ECOG PS scoring);
9. Expected survival ≥ 3 months;
10. Major organ function meeting the following criteria (no blood transfusions or blood products, and no medication correction within 2 weeks prior to treatment): Hematology: Absolute neutrophil count ≥ 1.5 × 10^9/L, platelet count > 80 × 10^9/L, hemoglobin ≥ 90 g/L; Biochemistry: Serum albumin ≥ 28 g/L, Thyroid-stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, free triiodothyronine (FT3) and free thyroxine (FT4) levels should also be checked. If FT3 and FT4 levels are normal, the patient can be included); Bilirubin ≤ 1.5 × ULN (7 days before first dose); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3 × ULN (7 days before first dose); Alkaline phosphatase (AKP) ≤ 2.5 × ULN; Serum creatinine ≤ 1.5 × ULN;
11. Women of childbearing potential: Must agree to use effective contraception or abstain from heterosexual intercourse from signing the informed consent form until at least 120 days after the last dose of the study drug. A negative serum human chorionic gonadotropin (HCG) test within one week prior to enrollment is required, and the patient must not be breastfeeding. Women who are menstruating, have not reached menopause (defined as ≥ 12 months of amenorrhea without other causes), and have not undergone sterilization procedures (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) are considered to be of childbearing potential;
12. For male participants with partners of childbearing potential, they must agree to use effective contraception or abstain from heterosexual intercourse from signing the informed consent form until at least 120 days after the last dose of the study drug. During this period, male participants must also agree not to donate sperm.

Exclusion Criteria:

1. Significant clinical bleeding symptoms or clear gastrointestinal bleeding tendencies (e.g., severe esophageal or gastric varices, active gastrointestinal ulcers, or vasculitis) within 3 months before enrollment. If fecal occult blood is positive during screening, a recheck is required, and if still positive, gastroscopy must be performed.
2. Active autoimmune diseases or history of autoimmune diseases with potential for recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, and hypothyroidism - only subjects controlled by hormone replacement therapy are allowed). Subjects with skin conditions requiring no systemic treatment (e.g., vitiligo, psoriasis, alopecia), childhood asthma fully resolved, and no intervention needed in adulthood may be included. Asthma patients requiring bronchodilators for medical intervention cannot be included.
3. Use of immunosuppressants or systemic steroids within 2 weeks before enrollment for immunosuppressive purposes (dose >10mg/day of prednisone or equivalent).
4. Allergy to any monoclonal antibodies, anti-angiogenesis targeted drugs, or excipients.
5. Known history of central nervous system metastases or hepatic encephalopathy.
6. Patients who are preparing for or have previously received organ or allogeneic bone marrow transplants.
7. Ascites with clinical symptoms requiring paracentesis or drainage, or ascites that has been drained within the past 3 months. Excludes asymptomatic ascites with minimal amounts seen on imaging.
8. Uncontrolled hypertension despite antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (average of ≥2 measurements). Previous hypertension crisis or hypertensive encephalopathy.
9. Severe iodine contrast allergy that prevents TACE treatment.
10. HBV-DNA >2000 IU/ml (or 10^4/ml); or HCV-RNA >10^3/ml; or HBsAg+ anti-HCV antibody positive patients.
11. Coagulation dysfunction (International normalized ratio (INR) >2.0, Prothrombin time (PT) >16s), bleeding tendencies, or receiving thrombolytic or anticoagulant therapy. Preventive use of low-dose aspirin and low molecular weight heparin is allowed.
12. Arterial thromboembolism events within the past 6 months, such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhage, cerebral infarction), or CTCAE grade 3 or higher deep vein thrombosis or pulmonary embolism.
13. Known hereditary or acquired bleeding and thrombosis disorders (e.g., hemophilia, coagulation disorders, thrombocytopenia).
14. Urinalysis indicating proteinuria ≥++ or 24-hour urine protein >1.0g.
15. Active infection, unexplained fever ≥38.5°C within 1 week before enrollment, or leukocyte count >15×10^9/L during screening. Therapeutic antibiotics within 2 weeks before enrollment (excluding prophylactic antibiotics administered intravenously for ≤48 hours).
16. Congenital or acquired immunodeficiencies (e.g., HIV infection).
17. History of other malignancies within the past 3 years (except for cured basal cell carcinoma and cervical carcinoma in situ).
18. Uncontrolled cardiac symptoms or diseases, such as NYHA class II or higher heart failure, or echocardiography showing left ventricular ejection fraction (LVEF) <50%; unstable angina; myocardial infarction within the past year; significant clinical supraventricular or ventricular arrhythmias requiring treatment or intervention on ECG; QTc >450ms (male) or QTc >470ms (female) on resting ECG.
19. Palliative radiotherapy within 4 weeks before enrollment, with radiotherapy area exceeding 5% of bone marrow area in bone metastasis patients.
20. Major vascular events (e.g., aneurysms requiring surgical repair or recent peripheral arterial thrombosis) within 6 months before enrollment.
21. Administration of live vaccines within 4 weeks before the study drug or potential live vaccine administration during the study.
22. Previous treatment with other anti-PD-1 antibodies or other PD-1/PD-L1 targeted immunotherapy, or previous targeted therapy.
23. Pregnant, breastfeeding women, or women of childbearing age unwilling to use contraception.
24. Any other factors that may affect study results or lead to study discontinuation, as judged by the investigator, such as alcoholism, drug abuse, other severe diseases requiring concurrent treatment (including psychiatric disorders), severe laboratory abnormalities, or family or social factors affecting patient safety.
25. Severe, non-healing or open wounds, active ulcers, or untreated fractures.
26. Major surgery within 4 weeks before enrollment (excluding diagnostic procedures) or expected need for major surgery during the study.
27. Use of strong CYP3A4/CYP2C19 inducers (e.g., rifampicin and similar agents) or strong CYP3A4/CYP2C19 inhibitors within 14 days before enrollment.
28. Participation in other drug clinical trials within 4 weeks before enrollment.
29. Other factors that the investigator deems unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Generally, the ORR is assessed for each participant every two treatment cycles(each cycle is 3 weeks).
  The ORR is defined as the proportion of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Generally, the DCR is assessed for each participant every two treatment cycles(each cycle is 3 weeks).
  The percentage of participants who achieve a BOR of CR, PR, or SD lasting at least 6 weeks, assessed according to RECIST 1.1 and mRECIST criteria.
Duration of response (DoR) | Generally, the DoR is assessed for each participant every two treatment cycles(each cycle is 3 weeks).
  DoR is defined as the time from the first recorded objective response (assessed according to RECIST 1.1 and mRECIST criteria) to the first recorded progression of target tumors (assessed according to RECIST 1.1 or mRECIST criteria) or to the date of any earlier death for any reason.
Progression-Free Survival (PFS) | Record the progression-freesurvival state of each participant at six months and twelve months after receiving the initial treatment.
  PFS is defined as the time from the first study treatment date to the first recorded tumor progression (according to RECIST 1.1 or mRECIST criteria, regardless of whether the study is still ongoing) or to the time of any earlier death for any reason.
Overall Survival (OS) | Record the survival state of each participant at six months and twelve months after receiving the initial treatment.
  OS is defined as the time from the first study treatment date to death from any cause.

OTHER OUTCOMES:
Number of peripheral blood lymphocytes | Peripheral blood lymphocyte will be conducted on Day 1±7 days before each of the first three cycles (each cycle is 3 weeks); thereafter, it will be checked every 6 weeks on Day 1±7 days until treatment end/withdrawal(no more than 12 months in total).
  To understand the changes in peripheral blood lymphocytes before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zheng, Principal Investigator
Locations (1):
- The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Result] Birkett MA, Day SJ. Internal pilot studies for estimating sample size. Stat Med. 1994 Dec 15-30;13(23-24):2455-63. doi: 10.1002/sim.4780132309. PMID 7701146
- [Result] Marshall E. Gene therapy death prompts review of adenovirus vector. Science. 1999 Dec 17;286(5448):2244-5. doi: 10.1126/science.286.5448.2244. No abstract available. PMID 10636774
- [Result] Yi L, Ning Z, Xu L, Shen Y, Zhu X, Yu W, Xie J, Meng Z. The combination treatment of oncolytic adenovirus H101 with nivolumab for refractory advanced hepatocellular carcinoma: an open-label, single-arm, pilot study. ESMO Open. 2024 Feb;9(2):102239. doi: 10.1016/j.esmoop.2024.102239. Epub 2024 Feb 6. PMID 38325225
- [Result] Lin XJ, Li QJ, Lao XM, Yang H, Li SP. Transarterial injection of recombinant human type-5 adenovirus H101 in combination with transarterial chemoembolization (TACE) improves overall and progressive-free survival in unresectable hepatocellular carcinoma (HCC). BMC Cancer. 2015 Oct 15;15:707. doi: 10.1186/s12885-015-1715-x. PMID 26470869
- [Result] Sivanandam V, LaRocca CJ, Chen NG, Fong Y, Warner SG. Oncolytic Viruses and Immune Checkpoint Inhibition: The Best of Both Worlds. Mol Ther Oncolytics. 2019 Apr 25;13:93-106. doi: 10.1016/j.omto.2019.04.003. eCollection 2019 Jun 28. PMID 31080879
- [Result] Ribas A, Dummer R, Puzanov I, VanderWalde A, Andtbacka RHI, Michielin O, Olszanski AJ, Malvehy J, Cebon J, Fernandez E, Kirkwood JM, Gajewski TF, Chen L, Gorski KS, Anderson AA, Diede SJ, Lassman ME, Gansert J, Hodi FS, Long GV. Oncolytic Virotherapy Promotes Intratumoral T Cell Infiltration and Improves Anti-PD-1 Immunotherapy. Cell. 2017 Sep 7;170(6):1109-1119.e10. doi: 10.1016/j.cell.2017.08.027. PMID 28886381
- [Result] Sharma P, Hu-Lieskovan S, Wargo JA, Ribas A. Primary, Adaptive, and Acquired Resistance to Cancer Immunotherapy. Cell. 2017 Feb 9;168(4):707-723. doi: 10.1016/j.cell.2017.01.017. PMID 28187290
- [Result] Qin S, Chan SL, Gu S, Bai Y, Ren Z, Lin X, Chen Z, Jia W, Jin Y, Guo Y, Hu X, Meng Z, Liang J, Cheng Y, Xiong J, Ren H, Yang F, Li W, Chen Y, Zeng Y, Sultanbaev A, Pazgan-Simon M, Pisetska M, Melisi D, Ponomarenko D, Osypchuk Y, Sinielnikov I, Yang TS, Liang X, Chen C, Wang L, Cheng AL, Kaseb A, Vogel A; CARES-310 Study Group. Camrelizumab plus rivoceranib versus sorafenib as first-line therapy for unresectable hepatocellular carcinoma (CARES-310): a randomised, open-label, international phase 3 study. Lancet. 2023 Sep 30;402(10408):1133-1146. doi: 10.1016/S0140-6736(23)00961-3. Epub 2023 Jul 24. PMID 37499670
- [Result] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971
- [Result] Galle PR, Finn RS, Qin S, Ikeda M, Zhu AX, Kim TY, Kudo M, Breder V, Merle P, Kaseb A, Li D, Mulla S, Verret W, Xu DZ, Hernandez S, Ding B, Liu J, Huang C, Lim HY, Cheng AL, Ducreux M. Patient-reported outcomes with atezolizumab plus bevacizumab versus sorafenib in patients with unresectable hepatocellular carcinoma (IMbrave150): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Jul;22(7):991-1001. doi: 10.1016/S1470-2045(21)00151-0. Epub 2021 May 27. PMID 34051880
- [Result] Tian L, Goldstein A, Wang H, Ching Lo H, Sun Kim I, Welte T, Sheng K, Dobrolecki LE, Zhang X, Putluri N, Phung TL, Mani SA, Stossi F, Sreekumar A, Mancini MA, Decker WK, Zong C, Lewis MT, Zhang XH. Mutual regulation of tumour vessel normalization and immunostimulatory reprogramming. Nature. 2017 Apr 13;544(7649):250-254. doi: 10.1038/nature21724. Epub 2017 Apr 3. PMID 28371798
- [Result] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Result] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Result] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Result] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Yang JD, Hainaut P, Gores GJ, Amadou A, Plymoth A, Roberts LR. A global view of hepatocellular carcinoma: trends, risk, prevention and management. Nat Rev Gastroenterol Hepatol. 2019 Oct;16(10):589-604. doi: 10.1038/s41575-019-0186-y. Epub 2019 Aug 22. PMID 31439937